CLINICAL TRIAL: NCT05186935
Title: A Multi-center, Pivotal, Non-randomized, Prospective, Open-label Study to Evaluate the Safety and Performance of the Hy2Care Injectable Hydrogel for the Repair of Cartilage Defects in the Knee
Brief Title: Advanced Cartilage Treatment With Injectable-hydrogel Validation of the Effect
Acronym: ACTIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hy2Care BV (Industry)
Collaborators: Avania (Industry); UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19019-Hy2Care-CIP01
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Cartilage Damage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): This is a multi-center, pivotal, non-randomized, prospective, open-label clinical investigation.
  Interventions: Device: Injectable Hydrogel treatment

INTERVENTIONS:
Device: Injectable Hydrogel treatment — The Injectable Hydrogel is a single use two-component injectable and bioresorbable hydrogel intended for treatment of cartilage defects in the knee, it is a medical device, exclusively for clinical investigations. The hydrogel is mixed intraoperatively and with an open knee procedure inserted into the cartilage defect, where it crosslinks and adheres to the cartilage with the use of a primer, allowing it to stay in place during movements of the knee. The hydrogel covers the defect to prevent formation of scar tissue and to allow cartilage to regenerate. The Injectable Hydrogel will be used in combination with general instruments typically used. The different components of the Injectable Hydrogel are arranged in two boxes: Components of the Injectable Hydrogel are grouped in plastic cover bags or packaged in vial boxes.This is a performance study, with a single arm, i.e Injectable Hydrogel. Recovery is monitored.

SUMMARY:
Multicentre, pivotal, non-randomized, prospective, open-label clinical investigation involving a new hydrogel, Hy2Care Injectable hydrogel, developed by Hy2Care B.V., Enschede, The Netherlands (hereafter referred to as "Hy2Care") to treat cartilage defects (< 2 cm2) in the human knee. The product aims at functional repair of cartilage defects in the knee and regeneration of cartilage.

The objective of this clinical investigation is to demonstrate the clinical safety and performance of the Hy2Care Injectable hydrogel. Data from this clinical investigation will be used to support a CE marking application for the Hy2Care Injectable hydrogel.

Sites will be selected based on a documented site qualification procedure. The Principal Investigator at each site will be selected based on confirmed expertise in the orthopaedic field. Each site will have a designated Principal Investigator and one or more study coordinators collectively responsible for the study data collection, inclusive of screening, enrolment, evaluation and documentation, in accordance with the International Organization for Standardization (ISO) 14155 guidelines for Good Clinical Practice. Per site, one physician will be assigned as Principal Investigator. Other physicians will be referred to as 'sub-investigators'.

DETAILED DESCRIPTION:
This is a multi-center, pivotal, non-randomized, prospective, open-label clinical investigation.

Safety oversight throughout will be provided by an independent Data Monitoring Committee (DMC) comprised of a clinical expert (knee surgeon), medical monitor and a senior statistician.

The clinical investigation will be split into two cohorts:

Safety cohort: The safety cohort is intended to determine the primary safety of the investigational device. In this cohort, 10 subjects will be treated at preferably 1 site. The safety cohort will receive the investigational device intraoperatively.

Following implantation of the investigational device in the initial safety cohort, the DMC will continuously monitor all emerging safety issues against the defined stopping rules of the clinical investigation. Any treatment-emergent severe adverse events or other safety concerns during the safety phase of the clinical investigation will immediately be referred, on a case by case basis, to the DMC for review against the stopping rules.

A formal review of safety against the stopping rules will be undertaken by the DMC when all of the safety cohort patients reach 3 months post- surgery. Subjects will be followed post-operatively for 12 months. The subjects in the safety cohort will undergo the same procedures as in the performance cohort, therefore all data acquired for the safety cohort will also be used to measure the performance and safety endpoints defined for the performance cohort.

Performance cohort: The performance cohort is intended to demonstrate the safety and performance of the investigational device. This cohort will be initiated after the completion of the safety phase and approval from the DMC. In the performance cohort 36 subjects will be treated at up to 5 investigational sites, where they will receive the investigational device intraoperatively.

The sample size has been calculated based on a minimal clinically important change (MIC) of 10 points in the composite Knee Injury and Osteoarthritis Outcome Score (KOOS, a patient reported outcome measure), compared to baseline, to provide an assessment of the performance of the investigational device. The primary endpoint is at 12 months follow-up. All subjects will be followed post-operatively for 12 months. Additional assessments occur at 1 month, 3 months and 6 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years and maximum 50 years of age at time of surgery;
2. Subject presents with a symptomatic defect in the knee with an NRS pain score of 4 or more;
3. Subject presents with defects in the knee cartilage with ICRS classification grades IIIa or IIIb;
4. Subject has a contained lesion of between 0.5 - 2 cm2 in size, and it is localized on the femoral condyle or trochlea;
5. Subject has an intact (ICRS grade ≤ 1) articulating joint surface (without "kissing lesions");
6. Subject is willing and able to comply with all aspects of the treatment, including MRI, after-care rehabilitation and evaluation schedule over a 12-month duration; and
7. Subject is willing and able to provide documented Ethics Committee-approved informed consent prior to initiation of any study procedures.

Exclusion Criteria:

1. Subject has a BMI > 30 kg/m2;
2. Subject has multiple defects to be treated that are interconnected or that have less than 0.5 cm of space in between them;
3. Subject underwent index-knee surgery < 3 months prior to study treatment.
4. Subject suffers from any medical condition that would hinder cartilage repair, such as additional unresolved comorbidities related to the index knee:

   1. Untreated anterior cruciate ligament (ACL) and/or posterior cruciate ligament (PCL) deficiency or,
   2. Complex ligamentous instability of the knee/ insufficient ligament support,
   3. Meniscus lesions, total or partial (more than 1/2 of total volume) resected meniscus,
   4. Limited joint mobility,
   5. Varus/valgus joint malalignment of more than 3 degrees,
   6. Subject has a trochlear cartilage defect that is associated with (suspected) patella maltracking without surgical correction,
   7. Subject underwent previous (failed) cartilage repair procedure(s), such as microfracture (MF), Osteochondral Autograft Transplantation (OATS) or Autologous Chondrocyte Implantation (ACI) with or without use of a scaffold (matrix) in the index knee.

   Comorbidities that are resolved during the same surgical procedure as the investigational device treatment, do not qualify for this exclusion criterion.
5. Subject has (history of) generalized osteoarthritis, defined as Kellgren-Lawrence grade >1 as determined from recent (<6 months at time of enrollment) X-ray;
6. Subject suffers from inflammatory joint diseases (e.g. rheumatoid arthritis, Bechterew disease, chondromatosis);
7. Subjects suffers from autoimmune disease, vascular or neurological disease;
8. Subject suffers from an active or recent local or systematic infection, or has a history of knee infections;
9. Subject has an active malignant tumor at the time of treatment;
10. Subject has hypersensitivity or allergy to the constituents of the product.
11. Pregnant or lactating women at the time of enrollment or women who are planning to become pregnant during the duration of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Performance | 12 months follow up
  Change from baseline in the composite (average of the 5 subscales) Knee Injury and OsteoArthritis Outcome Score (KOOS) at 12 months post-surgery.
  Performance:
  • Change from baseline in the composite (average of the 5 subscales) Knee Injury and OsteoArthritis Outcome Score (KOOS), at 12 months post-surgery.
  Hypothesis: Average change from baseline in the composite Knee Injury and OsteoArthritis Outcome Score (KOOS) at 12 months post-surgery with Hy2Care Injectable hydrogel is greater than a minimal clinically important change (MIC) of 10.

SECONDARY OUTCOMES:
Cartilage Regeneration via Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) | 12 months
  Determine the Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) II score at 12 months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Roel Custers, Dr, Principal Investigator — UMCU - Academic Hospital Utrecht; Barbara Kalkman, Dr, Study Director — UMCU - Academica Hospital Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No